CLINICAL TRIAL: NCT01757496
Title: Cough Assist in RSV-bronchiolitis
Brief Title: Cough Assist in Bronchiolitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with patient inclusion
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Principal Investigator, Stijn Verhulst, MD, PhD, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UZA-11/44/334
Record Dates: First submitted 2012-12-18; First posted 2012-12-31 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Bronchiolitis; Respiratory Syncytial Virus
Keywords: Bronchiolitis; Respiratory Syncytial Virus; Cough Assist; Physiotherapy
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cough Assist (Experimental): These children will receive 2 Cough Assist sessions daily.
  Interventions: Device: Cough Assist
- Control group (No Intervention): These children receive standard care but no physiotherapy.

INTERVENTIONS:
Device: Cough Assist
  Other Names: Philips-Respironics Cough Assist E70
  Arms: Cough Assist

SUMMARY:
RSV bronchiolitis in children is still associated with significant morbidity and mortality. RSV infection results in increased mucus production, edema and inflammation at the lower airways and impaired mucociliary clearance. Infants and children under the age of 1 year are particularly vulnerable to complications such as atelectasis and secondary bacterial infection. These children often need non-invasive or invasive ventilation. Atelectasis is common in these children because of smaller airways and decreased cough strength. There is still much uncertainty about the treatment of RSV. Treatment consists primarily of supportive therapy such as tube feeding and additional respiratory support if necessary. There is also limited evidence about the use of nebulizers with beta-agonists and/or hypertonic saline.

The cough assist is a mechanical in- and exsufflator used primarily in patients with neuromuscular diseases to augment cough capacity. In these patients, it was demonstrated that the use of assisted cough resulted in a significant decrease in the number of respiratory infections. Moreover, there is evidence that when used in the case of an acute respiratory deterioration such a massive atelectasis, the atelectasis can be corrected and intubation can be avoided. The aim of this study is to investigate if the use of the CoughAssist device in children with RSV bronchiolitis is associated with a better respiratory outcome.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 18 months admitted to our hospital with a clinical diagnosis of bronchiolitis in the RSV season or with a positive nasopharyngeal aspirate for RSV.

Exclusion Criteria:

* Children with congenital cardiac disease.
* Children with cystic fibrosis.
* Children with reactive airways disease.
* Children with neurological impairment including cerebral palsy.
* Children with neuromuscular disease.
* Children with upper GI surgery.
* Children with emphysema.
* Children with a known susceptibility to pneumothorax or with a pneumothorax in the past.

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Estimated)
Dates: Start 2012-09; Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Oxygen requirement | This will be investigated daily during hospitalization. The duration of hospitalization is estimated to 5-7 days.
  Number of days needing additional oxygen requirement

SECONDARY OUTCOMES:
Atelectasis | This will be investigated daily during hospitalization. The duration of hospitalization is estimated to 5-7 days.
  Development of atelectasis
Bronchoscopy | This will be investigated daily during hospitalization. The duration of hospitalization is estimated to 5-7 days.
  Need for bronchoscopy
Hypercapnia | This will be investigated daily during hospitalization. The duration of hospitalization is estimated to 5-7 days.
  Duration of hypercapnia
Hospitalization length | This will be determined at the moment of discharge. Average hospitalization length is estimated to be 5-7 days.
  Hospitalization length

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Verhulst, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (2):
- Belgium (2):
  - Antwerp University Hospital, Edegem
  - GZA Sint-Augustinus, Wilrijk